CLINICAL TRIAL: NCT04969887
Title: Ipilimumab and Nivolumab Combination Therapy in Patients With Selected Immunotherapy Sensitive Advanced Rare Cancers
Brief Title: Combination Immunotherapy in Rare Cancers Under InvesTigation
Acronym: MOST-CIRCUIT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONJ2021-002; CA209-6D6 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2021-07-06; First posted 2021-07-21 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Advanced Biliary Tract Cancer; Neuroendocrine Tumors; Female Reproductive System Neoplasm; MSI-H Solid Malignant Tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Genital Neoplasms, Female | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Masking Description: This is an open label study, all patients receive the same treatment as per the protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ipilimumab and Nivolumab (Experimental): All Subjects will be treated with: Nivolumab at 3 mg/kg and ipilimumab at 1 mg/kg concurrently every 3 weeks for 4 doses followed by nivolumab only at 480mg every 4 weeks until progression (up to 2 years)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) is a key regulator of T cell activity. Ipilimumab is a CTLA-4 immune checkpoint inhibitor that blocks T-cell inhibitory signals induced by the CTLA-4 pathway, increasing the number of tumor reactive T effector cells which mobilize to mount a direct T-cell immune attack against tumor cells. CTLA-4 blockade can also reduce T regulatory cell function, which may lead to an increase in anti-tumor immune response.
  Other Names: YERVOY ®
Drug: Nivolumab — A fully human immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed cell death-1 (PD-1,PCD-1) with immune checkpoint inhibitory and antineoplastic activities. Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs (antigen presenting cells). This results in the activation of T-cells and cell-mediated immune responses against tumor cells or pathogens. Activated PD-1 negatively regulates T-cell activation and and plays a key role in in tumor evasion from host immunity.
  Other Names: Opdivo

SUMMARY:
The four tumour streams that will be studied in this protocol are based on immunotherapy sensitive rare cancers from CA209-538 which will be further investigated under this protocol and divided into four groups:

1. Neuroendocrine cancers: Atypical bronchial carcinoid, neuroendocrine carcinoma and Grade 3 NETs independent of primary site (SCLC excluded)
2. Biliary tract cancers: Intrahepatic cholangiocarcinoma and gallbladder carcinoma
3. Gynaecological malignancies: Ovarian clear cell carcinoma, uterine clear cell carcinoma, uterine/ovarian carcinosarcoma, uterine leiomyosarcoma and vaginal/vulva squamous cell carcinoma
4. Mismatch repair protein deficient (MSI-H) cancers (excluding colorectal carcinoma).

The role of immunotherapy is being defined in more common cancer types, however because of their rarity, the efficacy of immunotherapy for these cancers is poorly defined.

This protocol provides an important opportunity to establish whether the combination of nivolumab & ipilimumab has efficacy in these cancers.

DETAILED DESCRIPTION:
This is a phase 2 clinical trial of nivolumab combined with ipilimumab in immunotherapy sensitive rare cancers. This study will allow an evaluation of the clinical benefit, as measured by progression free survival (PFS) >6 months and overall survival (OS), provided by nivolumab combined with ipilimumab.

Study Rationale Clinically advanced rare cancers pose a significant clinical challenge because evidence based treatments are seldom available for patients suffering from these malignancies. Despite little evidence that shows clinical benefit, these patients are often treated with chemotherapeutic agents that are used in patients with more common malignancies that arise from the same anatomical site. Furthermore, because of small numbers, patients are often excluded from clinical trials with newer agents. CA209-538 examined this treatment combination in three 'baskets' of rare cancers: rare upper gastrointestinal, gynaecological and neuroendocrine cancers. The cancers on study all individually had an incidence of <2/100000/year. The cancer specific survival of patients diagnosed with a rare malignancy is significantly lower than with common cancers highlighting the need to improve management and treatment of rare cancer patients. Given the success of cancer immunotherapy with checkpoint regulators such as ipilimumab and nivolumab in a range of different cancer types, it was postulated that these agents could be beneficial in rare cancers and improve the overall outlook of patients with these conditions. CA209-538 enrolled 120 rare cancer patients on study, clinical benefit rate was >30% across all baskets, long term survival follow-up is underway.

This study will enrol 240 participants, across 4 cohorts with histotypes which demonstrated clinical benefit on CA209-538. All participants will receive ipilimumab and nivolumab as combination immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
2. Target Population

   * a) Histologically confirmed Neuroendocrine cancers: Atypical bronchial carcinoid, neuroendocrine carcinoma and Grade 3 NETs independent of primary site (SCLC excluded); Biliary Tract Cancers: Intrahepatic cholangiocarcinoma, gallbladder carcinoma; Gynaecological malignancies: Ovarian clear cell carcinoma, uterine clear cell carcinoma, uterine/ovarian carcinosarcoma, uterine leiomyosarcoma, vaginal/vulva squamous cell carcinoma; Mismatch repair protein deficient (MSI-H) cancers (excluding colorectal carcinoma)
   * Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
   * Prior systemic therapy (≤1) for advanced disease is permitted if it was completed at least 4 weeks prior to enrolment, and all related adverse events have either returned to baseline or stabilized or participants are not suitable for, or if declining established standard therapies. For MSI-H rare cancers and atypical bronchial carcinoid only, patients will be eligible independent of the number of prior lines of systemic treatment received as long as treatment has been completed at least 4 weeks prior to enrolment.
   * Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration.
   * Measurable disease by CT or MRI per RECIST 1.1 criteria
   * Tumour tissue from an unresectable or metastatic site of disease must be available for biomarker analyses.
   * Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization:

     * WBC (white blood cells) > or = to 2000/μL
     * Neutrophils > or = to 1500/μL
     * Platelets > or = to 100 x103/μL
     * Hemoglobin > 9.0 g/dL
     * Serum creatinine < or = to 1.5 x ULN or creatinine clearance (CrCl) 40 mL/min (using the Cockcroft-Gault formula)
     * AST/ALT (aspartate transaminase/alanine transaminase) < or = to 3 x ULN (in the event of metastatic liver disease, an exception to this upper limit may be accepted in consultation with the study physician).
     * Total Bilirubin < or = to 1.5 x ULN (Upper limit of normal) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL).
   * Subject Re-enrolment: This study permits the re-enrolment of a subject that has discontinued the study as a pre-treatment failure (i.e. subject has not been treated) after obtaining agreement from the medical monitor prior to re enrolling a subject. If re-enrolled, the subject must be re-consented.
3. Age and Reproductive Status

   * Men and women, > or = to 18 years of age
   * Women of childbearing potential (WOCBP) must use method(s) of contraception. WOCBP should therefore use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for Nivolumab to undergo five half lives) after the last dose of investigational drug.
   * Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
   * Women must not be breastfeeding
   * Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1 percent per year. Men that are sexually active with WOCBP must follow instructions for birth control when the half life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 90 days plus the time required for the investigational drug to undergo five half lives. The half life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. Given the blinded nature of the study, men who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half lives) after the last dose of investigational drug.
   * Women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile and azoospermic men do not require contraception.

Exclusion Criteria:

1. Target Disease Exceptions

   * Active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI except where contraindicated in which CT scan is acceptable) evidence of progression for at least 8 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. Cases should be discussed with the medical monitor. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
2. Medical History and Concurrent Diseases

   * Prior combination treatment directed against the PD-1/PDL1 (Programmed Death Ligand 1) axis (anti PD 1, anti PD-L1, anti PD L2), and anti CTLA 4 antibody. Prior monotherapy with these agents or other immune-stimulating/regulating agents is permitted.
   * Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
   * Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
   * Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
   * Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
3. Physical and Laboratory Test Findings

   * Any positive test result for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
   * Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
4. Allergies and Adverse Drug Reaction

   * History of allergy to study drug components.
   * History of severe hypersensitivity reaction to any monoclonal antibody.
5. Sex and Reproductive Status

   * WOCBP who are pregnant or breastfeeding
   * Women with a positive pregnancy test at enrolment or prior to administration of study medication.
6. Other Exclusion Criteria

   * Prisoners or subjects who are involuntarily incarcerated
   * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Confirm the clinical efficacy of ipi/nivo in rare cancer histotypes which have demonstrated to be responsive to the regimen in the CA209-538 study. | At 12 weeks following registration then as assessed by standard care until progression.
  Clinical benefit rate for whole population (CR (complete response)+PR (partial response) assessed by radiographic evidence in accordance with RECIST 1.1 criteria
Determine the proportion of participants with progression free survival at 6 months | Enrolment on study until 6 months.
  Progression-free survival based on clinical or radiographic evidence of progressive disease according to RECIST 1.1 criteria at 6 months.

SECONDARY OUTCOMES:
To confirm the overall survival of participants receiving ipi/nivo in rare cancer histotypes which have demonstrated to be responsive to the regimen | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Quantification of OS.
To confirm the progression free survival of participants receiving ipi/nivo in rare cancer histotypes which have demonstrated to be responsive to the regimen | From date of enrolment until the date of first documented progression up to 5 years.
  Quantification of PFS
Quantification of treatment related toxicities to ipi/nivo according to CTCAE V5.0 | From 1st dose until 30 days following last dose [up to max 2 years + 30 days].
  Quantification of treatment related toxicities according to CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, MD, Study Chair — ONJCRI and Austin Health; Jonathan Cebon, MD, Study Chair — ONJCRI and Austin Health
Locations (18):
- Australia (17):
  - Border Medical Oncology Unit, Albury, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Cairns and Hinterland Hospital and Health Service, Cairns, Queensland
  - Townsville Hospital and Health Service, Douglas, Queensland
  - Townville Hospital and Health Service, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Bendigo Health Services, Bendigo, Victoria
  - Peninsula Health, Frankston, Victoria
  - Barwon Health, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCalllum Cancer Centre, Parkville, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - South West Healthcare, Warrnambool, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Derived] Carlino MS, Gao B, Michael M, Marshall H, Gunjur A, Chan H, Zielinski R, So J, Harris SJ, Kee D, Collins IM, Lam WS, Lyle M, Underhill C, Brown MP, Harrup R, Wong SF, Grady J, Ballinger M, Tavancheh E, Thomas DM, Palmer J, Wilkie K, Cebon J, Klein O. Nivolumab and Ipilimumab in Advanced Mismatch Repair-Deficient/Microsatellite Instability-High Noncolorectal Cancers: A Nonrandomized Clinical Trial. JAMA Oncol. 2025 Nov 13:e254721. doi: 10.1001/jamaoncol.2025.4721. Online ahead of print. PMID 41231502
- [Derived] Gao B, Carlino MS, Michael M, Underhill C, Marshall H, Gunjur A, So J, Kee D, Antill Y, Lam WS, Chan H, Harrup R, Hamilton A, Grady J, Ballinger M, Tavancheh E, Yoon WH, Palmer J, Thomas D, Wilkie K, Cebon J, Klein O. Nivolumab and Ipilimumab Combination Treatment in Advanced Ovarian and Endometrial Clear Cell Cancers: A Nonrandomized Clinical Trial. JAMA Oncol. 2025 Sep 1;11(9):982-989. doi: 10.1001/jamaoncol.2025.1916. PMID 40608313